CLINICAL TRIAL: NCT02801708
Title: Enhanced Detection of Underlying, Covert ATrial Fibrillation Using 7-day Holter Electrocardiogram in Patients With Embolic Stroke of Undetermined Source
Acronym: EDUCATE-ESUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Yuichi Miyazaki, Principal Investigator, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: NCVC-M27-017
Record Dates: First submitted 2016-06-04; First posted 2016-06-16 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Stroke
Keywords: Embolic stroke of undetermined source; Atrial fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine the diagnostic yield of continuous 7-day Holter ECG for detecting covert paroxysmal atrial fibrillation in patients with recent embolic stroke or transient ischemic attack (TIA) of undetermined cause after completion of a standard clinical work up including an initial 24-hour Holter monitoring.

DETAILED DESCRIPTION:
Covert atrial fibrillation (AF) is a relevant potential cause of a recently proposed clinical construct, "Embolic Stroke of Undetermined Source (ESUS)". However, routine post-stroke work up including 24-hour Holter monitoring may fail to detect paroxysmal AF. A recent systematic review has shown an increased AF detection rate with longer monitoring durations. The aim of this study is to evaluate the effectiveness of a novel ambulatory 7-day Holter ECG (EV-201, Parama-Tech inc.) for detecting AF in patients with recent ESUS after completion of a standard clinical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Recent ESUS (within 3 months of onset) defined as:

   A. Recent ischemic stroke (including transient ischemic attack with positive neuroimaging) visualized by brain imaging that is not lacunar B. Abscence of ≥ 50% stenosis or occlusion in cervical and intracranial arteries supplying ischemic area C. No atrial fibrillation after ≥ 24-hour Holter monitoring D. No intra-cardiac thrombus on transthoracic echocardiography E. No other major cardioembolic sources F. No other specific cause of stroke (for example, arteritis, dissection, migraine/vasospasm, drug abuse)
2. 20 years of age or older
3. Signed written informed consent

Exclusion Criteria:

1. Previously documented atrial fibrillation
2. Untreated hyperthyroidism
3. Pacemaker or implantable cardioverter defibrillator implanted or planned to implant
4. Estimated life expectancy < 12 months
5. Examination of seven-day Holter ECG not applicable within 3 months after stroke onset.
6. Patients considered inappropriate to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent embolic stroke of undetermined source
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Detection of any atrial fibrillation | After examination of 7-day Holter monitoring (within 90 days of stroke onset)

SECONDARY OUTCOMES:
Change of antithrombotic drugs | After the examination of 7-day Holter monitoring
Any ischemic or hemorrhagic event | 365 days after index stroke
Any adverse event related to 7-day Holter monitoring | After the examination of 7-day Holter monitoring
Time to detection of atrial fibrillation on 7-day Holter monitoring | After the examination of 7-day Holter monitoring
Atrial fibrillation burden | After the examination of 7-day Holter monitoring
  defined as the total time in atrial fibrillation devided by the total monitored time

CONTACTS AND LOCATIONS:
Overall Officials: Yuichi Miyazaki, MD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Derived] Miyazaki Y, Toyoda K, Iguchi Y, Hirano T, Metoki N, Tomoda M, Shiozawa M, Koge J, Okada Y, Terasawa Y, Kikuno M, Okano H, Hagii J, Nakajima M, Komatsu T, Yasaka M. Atrial Fibrillation After Ischemic Stroke Detected by Chest Strap-Style 7-Day Holter Monitoring and the Risk Predictors: EDUCATE-ESUS. J Atheroscler Thromb. 2021 May 1;28(5):544-554. doi: 10.5551/jat.58420. Epub 2020 Aug 15. PMID 32801289